CLINICAL TRIAL: NCT04428866
Title: Mechanisms of Post-Bariatric Hypoglycemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Joslin Diabetes Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000074
Record Dates: First submitted 2019-11-14; First posted 2020-06-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hypoglycemia
Keywords: Post-Bariatric Hypoglycemia; Roux-en-Y gastric bypass; Bariatric Surgery; Hypoglycemic clamp; Hormones; Microbiome
MeSH Terms: conditions — Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine, and fecal samples will be stored for up to 5 years for future analyses. DNA will be stored for additional expanded genotyping. Fecal samples and /or cultures from them may be used for mouse transfer experiments in the future.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with post-bariatric hypoglycemia: Individuals with history of Roux-en-Y gastric bypass surgery, who have a history of hypoglycemia will be recruited from the Joslin Hypoglycemia Clinic.
  Interventions: Diagnostic Test: Continuous Glucose Monitoring; Diagnostic Test: activity monitor; Diagnostic Test: Mixed meal tolerance test; Diagnostic Test: Glucagon Sensitivity Testing; Diagnostic Test: Hypoglycemic Hyperinsulinemic Clamp; Diagnostic Test: analysis of fecal microbiome
- Asymptomatic participants with Roux-en-Y gastric bypass (RYGB): Individuals with history of RYGB, without a history of or symptoms of hypoglycemia will be recruited from local postoperative surgical clinics and from the community.
  Interventions: Diagnostic Test: Continuous Glucose Monitoring; Diagnostic Test: activity monitor; Diagnostic Test: Mixed meal tolerance test; Diagnostic Test: Glucagon Sensitivity Testing; Diagnostic Test: Hypoglycemic Hyperinsulinemic Clamp; Diagnostic Test: analysis of fecal microbiome
- Control group: Individuals without a history of bariatric surgery will be recruited by local advertisement.
  Interventions: Diagnostic Test: Continuous Glucose Monitoring; Diagnostic Test: activity monitor; Diagnostic Test: Mixed meal tolerance test; Diagnostic Test: Glucagon Sensitivity Testing; Diagnostic Test: Hypoglycemic Hyperinsulinemic Clamp; Diagnostic Test: analysis of fecal microbiome

INTERVENTIONS:
Diagnostic Test: Continuous Glucose Monitoring — A CGM sensor (Dexcom G4 or other professional version available at onset of study) will be placed during visit 1 in blinded (masked) mode, and will be worn for 10 days. Data will be analyzed to determine patterns of glucose during both day and night intervals.
Diagnostic Test: activity monitor — The activity monitor (Fitbit Charge 2) will be worn by participants for 10 days to assess activity, concurrent with CGM sensor wear.
Diagnostic Test: Mixed meal tolerance test — After an overnight fast, participants will be given a standard liquid mixed meal; blood samples will be collected at baseline (fasting) and at defined time points after a meal for metabolic and hormonal analyses.
  Other Names: meal test
Diagnostic Test: Glucagon Sensitivity Testing — After baseline blood sampling, glucagon will be administered by injection, and blood samples will be collected for analysis of glucose and hormone responses. This will allow us to assess whether sensitivity to glucagon is altered in PBH.
Diagnostic Test: Hypoglycemic Hyperinsulinemic Clamp — This test will assess hormonal responses to hypoglycemia. Participants will arrive after an overnight fast. After baseline blood sampling, an infusion of insulin and glucose will be started, and infusions will be adjusted to allow glucose levels to drop very gradually. Blood samples will be collected for measurement of hormonal responses to lowering of glucose. This test will allow us to determine whether secretion of hormones which counteract hypoglycemia (counterregulatory hormones) is reduced in patients with PBH as compared with other groups.
  Other Names: Hyperinsulinemic Hypoglycemic Clamp
Diagnostic Test: analysis of fecal microbiome — Participants will be asked to provide a fecal sample, collected at home, which will be analyzed to determine the types of bacteria present in the feces.

SUMMARY:
Post-bariatric hypoglycemia (PBH) is an increasingly recognized syndrome that is incompletely understood.

The purpose of this study is to increase our level of understanding by investigating mechanisms contributing to this condition.

Participation in this study will take place over four visits, which will include the following:

* Wearing of a continuous glucose monitoring device;
* Providing a stool sample (collected at home);
* Measuring glucose and hormone levels in response to a meal;
* Measuring glucose and hormone levels in response to an injection of glucagon;
* Measuring hormone levels while glucose levels are gradually lowered, and during a controlled period of a low glucose level (hypoglycemic clamp).

Investigators will test the hypothesis that counterregulatory hormone responses are impaired in individuals with PBH, and that differences in the intestinal bacteria (microbiome) may contribute to this condition.

DETAILED DESCRIPTION:
Bariatric surgery is increasingly recognized as a potent tool for the treatment of type 2 diabetes (T2D), yielding not only weight loss but also rapid improvements in glycemia allowing discontinuation of diabetes-related medication within days after surgery. However, along with this metabolic success comes an increased incidence of severe hypoglycemia (termed post-bariatric hypoglycemia; PBH) for a subset of individuals.

The goal of these studies is to identify physiological and molecular mechanisms that underlie PBH, to determine whether these changes also contribute to surgery-induced improvements in glucose regulation (homeostasis), and to define potential new therapeutic interventions for PBH.

Participation in this study will take place over four visits, which will include the following:

* Detailed history, physical exam, and laboratory testing to determine study eligibility
* Assessment of glucose patterns using a masked continuous glucose monitor;
* Analysis of a stool sample (collected at home);
* Measuring glucose and hormone levels in response to a meal;
* Measuring glucose and hormone levels in response to an injection of glucagon;
* Measuring hormone levels while glucose levels are gradually lowered, and during a controlled period of a low glucose level (hypoglycemic clamp).

Investigators will test the hypothesis that counterregulatory hormone responses are impaired in individuals with PBH, and that differences in the intestinal bacteria (microbiome) and hormones produced in response to a meal may contribute to this condition.

ELIGIBILITY:
Inclusion Criteria:

1. For PBH group only: Males or females diagnosed with ongoing post-bariatric hypoglycemia with prior episodes of neuroglycopenia, unresponsive to dietary intervention (low glycemic index, controlled carbohydrate portions) and trial of acarbose therapy at the maximally tolerated dose.
2. For post-RYGB group without PBH: Males or females with history of RYGB and no history of symptomatic hypoglycemia.
3. For non-surgical controls only: Males or females with no history of upper gastrointestinal surgery and no history of hypoglycemia or diabetes.
4. Age 18-70 years of age, inclusive, at screening.
5. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria:

1. Documented hypoglycemia occurring in the fasting state (> 12 hours fast);
2. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
3. Hepatic disease, including serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
4. Congestive heart failure, New York Heart Association class II, III or IV;
5. History of myocardial infarction, unstable angina or revascularization within the past 6 months or 2 or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use.
6. History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia
7. Concurrent administration of β-blocker therapy;
8. History of a cerebrovascular accident;
9. Seizure disorder (other than with suspect or documented hypoglycemia);
10. Active treatment with any diabetes medications except for acarbose;
11. Active malignancy, except basal cell or squamous cell skin cancers;
12. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
13. Known insulinoma;
14. Major surgical operation within 30 days prior to screening;
15. Hematocrit < 33% (women) or <36% (men);
16. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
17. Blood donation (1 pint of whole blood) within the past 2 months;
18. Active alcohol abuse or substance abuse;
19. Current administration of oral or parenteral corticosteroids;
20. Pregnancy and/ or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intrauterine device, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
21. Use of an investigational drug within 30 days prior to screening.

There will be no involvement of special vulnerable populations such as fetuses, neonates, pregnant women, children, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable populations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with post-bariatric hypoglycemia will be recruited from the the Joslin Hypoglycemia Clinic.
  Individuals who have had RYGB but have no symptoms of hypoglycemia will be recruited from local bariatric programs and via advertisement.
  Control individuals will be recruited via advertisement locally.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Metabolic responses during experimental hypoglycemia induced by hypoglycemic clamp and/or mixed meal testing | July 2023
  Metabolites will be measured at set time points after the start of insulin or mixed meal. For the hypoglycemic clamp, a time-trend analysis will be performed to identify the glucose level at which each metabolite rises significantly above the linear average of its preceding values. Linear mixed effects modeling will be utilized to identify group- and time-dependent differences in metabolite responses. Data will be checked to ensure variables conform to assumptions of the analysis. Sensitivity analysis will determine whether missing data are randomly associated with clinical or experimental phenotypes, and assess the impact of missing data on conclusions. Relationships between clinical and metabolic variables will be analyzed using Pearson correlation, and adjusted for multiple comparisons using Benjamini-Hochberg testing.
Hormonal responses during experimental hypoglycemia induced by hypoglycemic clamp and/or mixed meal testing | July 2023
  Counterregulatory hormones will be measured at set time points after the start of insulin or mixed meal. For the hypoglycemic clamp, a time-trend analysis will be performed to identify the glucose level at which each hormone rises significantly above the linear average of its preceding values. Linear mixed effects modeling will be utilized to identify group- and time-dependent differences in counterregulatory hormone responses. Data will be checked to ensure variables conform to assumptions of the analysis. Sensitivity analysis will determine whether missing data are randomly associated with clinical or experimental phenotypes, and assess the impact of missing data on conclusions. Relationships between clinical and hormonal variables will be analyzed using Pearson correlation, and adjusted for multiple comparisons using Benjamini-Hochberg testing.
Assessment of glucagon responsiveness during glucagon stimulation testing | July 2023
  Glucose response to glucagon will be assessed by measurement of glucose levels at baseline, and at set time points after glucagon injection. Linear mixed effects modeling will be utilized to identify group- and time-dependent differences in glucose response to glucagon. Relationships between clinical variables and glucose levels in response to glucagon will be analyzed using Pearson correlation, and adjusted for multiple comparisons using Benjamini-Hochberg testing.
Assessment of hormonal responses during glucagon stimulation testing | July 2023
  Hormonal response to glucagon will be assessed by measurement of hormone levels at baseline, and at a set time point after glucagon injection. Linear mixed effects modeling will be utilized to identify group- and time-dependent differences in hormonal response to glucagon. Relationships between clinical variables, glucose levels, and hormonal levels in response to glucagon will be analyzed using Pearson correlation, and adjusted for multiple comparisons using Benjamini-Hochberg testing.
Analysis of microbiome differences in patients with PBH | July 2023
  Microbiome will be characterized by sequencing to obtain metagenomic data and pathway analysis; all data will be adjusted for multiple comparisons.

SECONDARY OUTCOMES:
Correlation between counterregulatory hormone response to experimental hypoglycemia and magnitude of hypoglycemia as determined by continuous glucose monitoring (CGM) | July 2023
  CGM data will be analyzed to assess mean, median, peak, and nadir sensor glucose values, glycemic variability (GV), severity and length of hypoglycemia (% time glucose <70, <60, <54 mg/dL), and number and duration of severe hypoglycemia (sensor glucose <54, duration >15 minutes) will be quantified. Metrics will be assessed over 24 hours and during daytime (6 AM to midnight) and nighttime (midnight to 6 AM) independently. Magnitude of hypoglycemia will be correlated with counterregulatory hormone levels during experimental hypoglycemia.
Correlation between hypoglycemia frequency (as determined by CGM) and microbiome | July 2023
  Metagenomic data will be correlated with hypoglycemia frequency determined by CGM.
Correlation between hypoglycemia frequency (as determined by CGM) and counterregulatory hormones. | July 2023
  Hypoglycemia data (from CGM) will be correlated with counterregulatory hormone response to experimental hypoglycemia.

OTHER OUTCOMES:
Safety Outcome - Hyper - and hypoglycemia during the study. | July 2023
  Participants will be closely monitored and glucose levels will be checked regularly at set time points during study visits. Symptoms of hypoglycemia will also be assessed at set time points during visits, and as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elizabeth Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data may be shared with other researchers with permission of local institutional review boards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of study results
Access Criteria: Data will be shared with academic investigators with approval of local institutional review boards.

REFERENCES:
- See also: Joslin Diabetes Center: Mechanisms of PBH recruitment website with contact information — https://www.joslin.org/research/clinical-research/clinical-trials/mechanisms-post-bariatric-hypoglycemia